CLINICAL TRIAL: NCT01323140
Title: An Open Label, Dose-Proportionality, Bioavailability and Dose- Titration Investigation of the Pharmacokinetics, Metabolism, Efficacy and Safety of Two Testosterone Matrix Transdermal Systems (28 cm2 and 48 cm2) in Hypogonadal Men
Brief Title: Pharmacokinetics, Metabolism, Efficacy, and Safety Study of Two Testosterone Matrix Transdermal Systems
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TM1103
Record Dates: First submitted 2011-03-21; First posted 2011-03-25 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-11

CONDITIONS: Hypogonadism
Keywords: hypogonadism, testosterone, transdermal system
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMTS treatment (Experimental): Following a lead-in dose-proportionality phase (Days 1-2) and a site-to-site bioavailability phase (Days 2-9), subjects were dosed for efficacy analysis beginning on Day 9 at dose level B (a single 48 cm2 testosterone matrix transdermal system). Based on pharmacokinetic (PK) analysis of blood samples drawn on Day 16, on Day 22 subjects could be dose-titrated up to dose level C (one 28 cm2 plus one 48 cm2 TMTS), down to dose level A (one 28 cm2 TMTS), or remain at dose level B. Subjects at all dose levels were pooled for primary efficacy analysis on Days 29/30.
  Interventions: Drug: testosterone matrix transdermal system

INTERVENTIONS:
Drug: testosterone matrix transdermal system

SUMMARY:
Watson's testosterone transdermal system delivers male sex hormone through skin for the treatment of men with sex hormone insufficiency.

DETAILED DESCRIPTION:
The present study is designed to characterize efficacy and safety of testosterone from the Watson's testosterone matrix transdermal system (TMTS).

ELIGIBILITY:
Inclusion Criteria:

* Male, 18 - 65 years of age;
* Documented testosterone deficiency;
* BMI 18 to 33.

Exclusion Criteria:

* Evidence of prostate cancer and benign prostate hyperplasia;
* Taking medications that interfere testosterone metabolism;
* History of alcohol or drug substance abuse;
* Abnormal ECG;
* Allergic to transdermal products;
* Skin condition that interfere transdermal system application and assessment

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keshava Kumar, PhD, MHSA, Study Director — Watson Pharmaceuticals
Locations (2):
- United States (2):
  - Watson Investigational Site, Fort Meyers, Florida
  - Watson Investigational Site, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 40
Completed | 38
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.1 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With Testosterone Levels in the Normal Range.
Description: Testosterone serum concentration was determined on Day 29/30 and pharmacokinetic (PK) parameters including Cavg and Cmax were calculated for efficacy assessment. Acceptance was defined as at least 75% of subjects with Cavg in the normal range (>= 300 ng/dL to <= 1030 ng/dL), at least 85% of subjects with Cmax <= 1500 ng/dL, no more than 5% of subjects with Cmax between 1800 and 2500 ng/dL, and no subject with Cmax >= 2500 ng/dL.
Time Frame: Day 29/30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment: As specified in the Protocol, subjects were dose-titrated during treatment and subjects at all resulting dose levels were pooled for primary efficacy analysis. After dose-titration, 20 subjects were receiving TMTS at dose level B (one 48 cm2 TMTS) and 18 subjects were receiving TMTS at dose level C (one 48 cm2 and one 28 cm2 TMTS). See also Arm description.
Arm/Group | Treatment
Number analyzed (Participants) | 38
percentage of participants | 68.4 (132.9) [53.6 to 83.2]

ADVERSE EVENTS:
Time Frame: First test article administration to study exit.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 6/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=40)
Application site irritation (General disorders) | 3 (4)
Headache (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less